CLINICAL TRIAL: NCT04318756
Title: The Italian Version of the Cancer Worry Scale . A Pancreatic Context Adaptation and Reliability Analysis
Brief Title: The Italian Version of Cancer Worry Scale
Acronym: CWS_Ita
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: 2458 CWS
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-01

CONDITIONS: Cancer Fear; Pancreatic Cancer
Keywords: cancer worry scale; cancer fear; pancreatic cancer risk; pancreatic cancer
MeSH Terms: conditions — Pathophobia; Pancreatic Neoplasms | interventions — Protein Biosynthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Italian patients suffering from mucinous neoplasms: Italian patients suffering from mucinous neoplasms will follow a brief interview made by a psychologist. The interview of pilot group will be record to allow us to investigate and track detail that will highlight the comprehension of cancer worry scale and participants' suggestion. Moreover during the session will be ask to patients to fill inn Irritability-Depression-Anxiety Scale and Patient Health Questionnaire-9 to evaluate other psycho-emotional information about fear of cancer
  Interventions: Behavioral: Translation and cultural adaptation go the cancer worry scale
- Italian patients with familiarity/genetic predisposition: Italian patients with familiarity/genetic predisposition will follow a brief interview made by a psychologist. The interview of pilot group will be record to allow us to investigate and track detail that will highlight the comprehension of cancer worry scale and participants' suggestion. Moreover during the session will be ask to patients to fill inn Irritability-Depression-Anxiety Scale and Patient Health Questionnaire-9 to evaluate other psycho-emotional information about fear of cancer
  Interventions: Behavioral: Translation and cultural adaptation go the cancer worry scale

INTERVENTIONS:
Behavioral: Translation and cultural adaptation go the cancer worry scale — To develop and validate the Italian version of Cancer worry scale using high risk subjects for familiarity/genetic predisposition and patients with premalignant lesions.
  Other Names: 1) Preliminary pilot testing conducted on a pilot group on patients under surveillance for pancreatic cancer

SUMMARY:
An Italian language version of the Cancer Worry Scale is not available yet.

The aim of this study is to develop and validate the Italian version of Cancer Worry Scale through subjects at high risk of pancreatic cancer for familiarity/genetic predisposition, or suffering from premalignant cystic lesions.

DETAILED DESCRIPTION:
The Fear of Cancer remains a significant problem for subjects enrolled surveillance programs. This emotional condition can influence the patients' wellbeing and their adherence to treatments. No results coming from the application of Cancer Worry Scale on high-risk of Pancreatic cancer individuals have been provided yet.

The fear is an emotional reaction that can be the result of interpretation and cognitions of perceived internal cues and/or external cues. To objectify this emotion, a cancer worry scale, has been developed to investigate the fear in female breast cancer survivors. The proposed scale assesses the psychological distress caused by fear of cancer.

The detection of high level of fear can prevent problematic behaviours, including anxious preoccupation, avoidance, and excessive checking, and moreover it can help patients to reduce difficulties in performing the individual's daily and social activities. The scale could use to evaluate the psychological burden produced by the enrolment in a surveillance program due to a certain predisposition to Pancreatic cancer. One step forward will be to manage those individuals with high-level of Fear of cancer, providing them a proper psychological support.

At the General and Pancreatic Surgery Unit of the Pancreas Institute, some experimental self-made psychological support programs that investigate different psychologic distress through validated instruments, like anxiety, depression, perceived stress and global assessment or quality of life have been built up. It must be noted that the scale is not available specifically for Pancreatic cancer (originally it was created for breast cancer) , and for the Italian language, thus it has never been applied in an italian surveillance/follow-up program dealing with Pancreatic cancer. Nowadays, there is only a well-structured paper assessing psychological factors associated with cancer worries in high risk participants in a pancreatic cancer surveillance program. Differently than what has been already reported by Konings et al, the cohorts of patients that will be considered are heterogeneous, reflecting more accurately the real-life scenario of the subjects to whom the scale is administered to. In addition, this may help to identify those individuals that may benefit from a psychological support, in order to prevent a withdrawal from the surveillance program.

However, a cut-off has not been provided yet. With next step study we'll aim at determining a cut-off for the detection clinically relevant worry for cancer.

ELIGIBILITY:
Inclusion Criteria:

Subject will be recruited from the current outpatients' clinic activity of the General and Pancreatic Surgery Unit, Pancreas Institute, Verona University Hospital. Subjects must be able to read and write in Italian. After obtained informed consent we will ask them to participate to preliminary pilot phase.

The interview of the pilot group will be audio recorded to allow to investigate and track detail that will highlight the comprehension of scale and participants' suggestion.

Patients affected by cynic neoplasm (group A) and high risk subjects for familiarity/genetic predisposition (group B) are currently enrolled at General and Pancreatic Surgery Unit of the Pancreas Institute of the University of Verona.

Group A Patients with premalignant lesions (such as intraductal papillary mucinous neoplasms) that are followed-up at our Institution, to detect any clinic-radiological progression. Subjects older than 18 will be enrolled.

Group B

The enrolment criteria were the following :

* Having at least 45 years of age or 10 years younger than the age of the youngest relative with pancreatic cancer (only for subject with familiar history of pancreatic cancer)
* Having at least 40 years of age or 5 years younger than the age of the youngest relative with pancreatic cancer (only for subject with familial pancreatitis and subject affected by Lynch syndrome with at least one relative first- or second-degree affected by pancreatic cancer and subject having a known genetic mutation with at least a first-degree relative or a second-degree relative affected by pancreatic cancer
* Having at least 30 years of age for subject with Familial Multiple Melanoma Syndrome
* Having at least 30 years of age for patients affected by Peutz-Jeghers syndrome.

The interview of pilot group will be record to allow us to investigate and track detail that will highlight the comprehension of cancer worry scale and participants' suggestion.

Exclusion Criteria:

* patients who not meet eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject will be recruited from the current outpatients' clinic activity of the General and Pancreatic Surgery Unit, Pancreas Institute, Verona University Hospital. Subjects must be able to read and write in Italian. After obtained informed consent we will ask them to participate to preliminary pilot phase.
  The interview of the pilot group will be audio recorded to allow to investigate and track detail that will highlight the comprehension of scale and participants' suggestion.
  Patients affected by cynic neoplasm (group A) and high risk subjects for familiarity/genetic predisposition (group B) are currently enrolled at General and Pancreatic Surgery Unit of the Pancreas Institute of the University of Verona.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Syntactic and semantic equivalence of Cancer worry scale' items between English and Italian language and vice versa | 1 month
  the Syntactic and semantic equivalence of scale between two languages will be verified through the evaluation of differential item functioning analysis

SECONDARY OUTCOMES:
Face Validity of cancer worry scale on Italian subjects | 6 months
  Face Validity will be measured through the evaluation of Clarity/ comprehensibility of each item of cancer worry scale (format and meaning)
Exploratory comparison between Patients Health Questionnaire and Irritability Depression Anxiety Scale and cancer worry scale | 9 months
  the comparison will be done considering the total score of scales